CLINICAL TRIAL: NCT00171873
Title: Study to Investigate the Antiproliferative Effect of Octreotide in Patients With Metastasized Neuroendocrine Tumors of the Midgut
Brief Title: Antiproliferative Effect of Octreotide in Patients With Metastasized Neuroendocrine Tumors of the Midgut
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carmen Schade-Brittinger (Other)
Responsible Party: Sponsor-Investigator, Carmen Schade-Brittinger, Sponsor-representative, Philipps University Marburg
Organization: Philipps University Marburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSMS995ADE05; NCT00202085 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Tumors
Keywords: Double blind; Phase III; Disease; Clinical trial; Octreotide; Neuroendocrine tumor; Cancer; Tumor; Midgut
MeSH Terms: conditions — Neuroendocrine Tumors; Disease; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Octreotide LAR (Long Acting Release) (Experimental): Octreotide LAR 30 mg intramuscularly every 28 days
  Interventions: Drug: Octreotide LAR (Long-acting release)
- Placebo (Placebo Comparator): Placebo - Sodium chloride intramuscularly every 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide LAR (Long-acting release) — 30 mg intramuscularly every 28 days
  Other Names: SMS995
  Arms: Octreotide LAR (Long Acting Release)
Drug: Placebo — Sodium chloride intramuscularly every 28 days
  Arms: Placebo

SUMMARY:
Placebo-controlled prospective randomized phase III study to investigate the antiproliferative effect of octreotide in patients with metastasized neuroendocrine tumors of the midgut

ELIGIBILITY:
Inclusion Criteria:

* Therapy-naive patients with histologically confirmed diagnosis of a locally inoperable or metastasized well-differentiated neuroendocrine tumor of the midgut
* curative surgery impossible
* two-dimensional tumor formation assessable by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
* Age ≥ 18
* Karnofsky-index > 60
* written informed consent
* proliferation index for Ki67

Exclusion Criteria:

* hypersensitivity to octreotide
* poorly differentiated or small cell neuroendocrine tumors
* primary tumor outside of the midgut
* prior treatment with somatostatin-analogue > 4 weeks
* prior treatment with alpha-interferon, chemotherapy, or chemoembolisation
* participation in any other clinical trial
* pregnancy or lactation
* no secondary malignancy in anamnesis; with the exception of patients without any manifestation of the secondary malignancy (without relapse) after curative therapy within the last five years
* severe decompensated organ malfunction (heart-, liver- insufficiency)

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2001-09; Primary Completion 2008-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Arnold, MD, Prof, Principal Investigator — Philipps University Marburg
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München

REFERENCES:
- [Derived] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide LAR (SMS995): Octreotide LAR (Long-acting release) 30 mg intramuscularly every 28 days
Period: Overall Study
Arm/Group | Octreotide LAR (SMS995) | Placebo
Started | 42 | 43
Completed | 33 | 40
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 5 | 0
Not completed — Switched to Octreotide | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide LAR (SMS995) | Placebo | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Median (Full Range); unit: years] | 63.5 [38 to 79] | 61 [39 to 82] | 62 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression Documented by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
Description: Median time to tumor progression at the time of the planned interim analysis that includes all data observed until June 2008.
Time Frame: Up to 7 years
Population: Conservative Intent to Treat (ITT) population consisting of all participants who received study drug. 3 participants in the Octreotide group and 1 participant in the placebo group without liver involvement at the beginning of the study were excluded from this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Octreotide LAR (SMS995) | Placebo
Number analyzed (Participants) | 39 | 42
Months | 14.3 [11.0 to 28.8] | 6.0 [3.7 to 9.4]

2. Secondary Outcome: Objective Response Rates According to World Health Organization (WHO) Criteria at 3 Month Intervals
Time Frame: at 3 month intervals
Reporting Status: Not Posted

3. Secondary Outcome: Biochemical Response at 3 Month Intervals
Time Frame: at 3 month intervals up to 18 moths
Reporting Status: Not Posted

4. Secondary Outcome: Symptom Control at 3 Month Intervals
Time Frame: at 3 month intervals up to 18 moths
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life (Standardized Questionnaire) at Three-month Intervals in Comparison With the Start of the Study
Time Frame: at three-month intervals
Reporting Status: Not Posted

6. Secondary Outcome: Survival
Time Frame: at least on a monthly basis
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Octreotide LAR (SMS995) | Placebo
Serious Adverse Events (participants affected / at risk) | 11/42 | 10/43
Other Adverse Events (participants affected / at risk) | 19/42 | 11/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide LAR (SMS995) (N=42) | Placebo (N=43)
General Disorder (General disorders) | 11 | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide LAR (SMS995) (N=42) | Placebo (N=43)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 | 8
Hematopoietic system (Blood and lymphatic system disorders) | 5 | 1
General Health (General disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.